CLINICAL TRIAL: NCT02247271
Title: The Role and Effectiveness of Diabetes Coaches in British Columbia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Patrick T. McGowan, PhD, Professor, School of Public Health and Social Policy, University of Victoria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-775-Diabetes
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: peer coaches
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetes health coach support (Other): The intervention is that subjects will receive coach support once a week for 30 minutes for six months. Support is provided by a Diabetes Coach who uses self-management support strategies to assist subjects to achieve their personal health goals.
  Interventions: Behavioral: Diabetes health coach support

INTERVENTIONS:
Behavioral: Diabetes health coach support — Receives support from a trained peer health coach for a six month period

SUMMARY:
This project is a partnership between the University of Victoria and the eleven Diabetes Health Centres in the Fraser Health Region of British Columbia, Canada. The primary goal of this project is to evaluate the feasibility, viability, and effectiveness of using peer health coaches to assist persons with type 2 diabetes who are experiencing challenges in managing their diabetes. The University of Victoria will recruit and train sixty coaches with various cultural and socioeconomic backgrounds representing a community of practice. Coaches will also have type 2 diabetes or be familiar with type 2 diabetes and will have led or taken the Diabetes Self-Management Program in English, Punjabi or in Aboriginal communities. Training will also include navigating the health care system, accessing mandated health and employment- related services, importance of medication adherence and ability to understand health care instructions. One hundred and fifty subjects with type 2 diabetes will be recruited by Diabetes Health Educators or through community newspaper ads. Eligibility criteria for subjects include: adults with type 2 diabetes who speak English or Punjabi living in the Fraser Health region. A one group pre-post matched design will be used. Both participants and coaches will complete questionnaires at baseline, six and twelve months. The Diabetes Coaches will provide assistance to subjects for a period of 6 months. A project community advisory committee comprised of the researchers, Diabetes Centre administrative staff, clinicians, coaches, subjects, key community leaders and representatives from the diabetes industry will meet every three months to guide implementation and sustainability. Qualitative research methods (i.e., focus groups and interviews) will be used to gather feedback, perspectives, and opinions of all the stakeholders.

DETAILED DESCRIPTION:
SUBJECT RECRUITMENT. Recruitment will take place during the first year by Diabetes Centre Educators in the Fraser Health region and through community newspaper ads. In total, 150 subjects will be recruited, along with 60 coaches. Diabetes Centre Educators will refer interested clients who will be contacted by the study coordinator. Persons responding to community newspaper ads will contact the study coordinator directly. Interested subjects will receive a full description of the study and confirm that they want to register. A package containing the Fraser Health Consent Form and a set of questionnaires will be mailed to them.

DIABETES COACH RECRUITMENT AND TRAINING. Recruitment and training will occur in the first 6 months. Criteria includes: living in the Fraser Health Region, adults, having type 2 diabetes or living with someone who has type 2 diabetes, and having similar cultural and ethnic background as members of the community. The coaches will most likely have already completed participation in a self-management program and therefore be knowledgeable in using self-management support strategies.

Competency-based training will be conducted to alleviate potential health professional concerns regarding the quality of service provided by non-professionals. Based on the experience using health workers to assist patients with diabetes (14), our project will provide a six-week training which will include:

* self-management support strategies as per the Five As approach (15);
* the Training Curriculum for Health Coaches (16);
* using behavioural change strategies on exercise, eating habits, smoking, and alcohol use developed by the national Service's Health Trainer Manual (17);
* basic information on diabetes and associated chronic diseases;
* finding and using governmental and community services;
* navigating the health care system; and if required
* completing the Diabetes Self-Management Program. Health coaches will undergo a final exam to receive certification from the University of Victoria. Subjects will be paired with a diabetes coach by the study coordinator. An innovative aspect of the proposed research is that baseline outcome measures will be calculated and used to tailor the coach intervention. For example one of the measures, the Patient Activation Measure (18), assesses an individual's knowledge, skill and confidence in managing their health, and specifies the types of interventions to increase activation. This is important because a systematic review of evidence on the performance of the Patient Activation Measure conducted by the National Health Service in 2012 (19) found that: higher PAM scores were associated with increased patient participation, significantly better health and significantly lower rates of doctor office visits, emergency room visits, and hospital nights; healthy behaviours; improved adherence to treatment; and with better doctor-patient communication. The study is also using other outcome measures that enable the tailoring of the intervention, for example the medication adherence and health literacy measures.

The coach will work with the subject by telephone for six months. Coaches will help subjects gain the knowledge, skills, tools, and confidence they need to become active participants in their care so that they can reach their self-identified health goals. The coach will also assist the patient to participate in the Diabetes Self-Management Program, learn and use effective self-management strategies (i.e., action plans and problem solving); understand and follow their medication regimen; access community resources (e.g., recreation centre); and receive eligible federal and provincial mandated services (e.g., income assistance, disability benefits), and learn about and use community resources (e.g., recreation centres), and assist the patient to use mandated services (e.g., income assistance).

With respect to innovation, it is time to tap the (largely) untapped resource of peer support to deal with the burden of diabetes (20). According to the World Health Organization, patients and families are the most undervalued assets in the health care system (10). A potential solution is to train peers to " coach" or work collaboratively to deliver self-management support to persons with diabetes. Peer coaching is defined as " helping patients gain the knowledge, skills, tools, and confidence they need to become active participants in their care so that they can reach their self-identified health goals" (21). A peer coaching intervention complements, enhances, and increases the comprehensiveness of primary care services, while increasing patient centredness and reducing fragmentation of care (21). While family, caretakers, friends and healthcare professionals can fill the role of advisor, supporter and role model, they can rarely fulfill all three roles. Peer health coaches, however, can fulfill all three roles and also benefit personally. Utilizing peer advisors for chronic disease management and particularly for people with type 2 diabetes has the potential to be cost effective (22). In a systematic review of the literature on peer support for chronic and complex conditions, the authors found more evidence that peer self-management support was effective with socially disadvantaged groups. Improved health outcomes were found for a Bangladeshi and Maori community with culturally relevant peer support in diabetes programs (23).

ELIGIBILITY:
Inclusion Criteria:

* adults, living in Fraser Health Region of British Columbia, type 2 diabetes, ability to speak English or Punjabi

Exclusion Criteria:

* Type 1 diabetes

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09-01; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | one year
  This is a composite measure

SECONDARY OUTCOMES:
glycated hemoglobin test (A1C) | one year
  Measures blood glucose level
Diabetes Empowerment Scale (DES) | one year
  Assesses subjects' perception of empowerment to manage diabetes
Self-efficacy | one year
  Measures confidence in managing diabetes
Self-reported health | one year
  Assess subjects' perception of their health status
Fatigue | one year
  Assesses subjects' perception of fatigue level
Pain | one year
  Assesses subjects' perception of pain level
Patient Health Questionnaire (PHQ-9) Depression Scale | one year
  Assesses subjects' perception of depression experience
Communication with physician | one year
  Assesses' subjects' communication with their doctor
Medication Adherence scale | one year
  Measures subjects' adherence to prescribed medication
Chow 3 question health literacy scale | one year
  Measures health literacy
Self-reported healthcare utilization | one year
  Self-report number of doctor visits, emergency room visits, and nights in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T McGowan, PhD, Principal Investigator — University of Victoria
Locations (1):
- UVictoria, Delta, British Columbia, Canada

REFERENCES:
- See also: Study proposal citations — http://www.selfmanagementbc.ca/uploads/Common/References.pdf